CLINICAL TRIAL: NCT04529291
Title: InertiaLocoGraphy as a Biomarker of Immunoglobulin Therapy Efficacy in Chronic Inflammatory Demyelinating Polyradiculoneuropathy
Acronym: SW_CIDP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The IP decided to stop.
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SW_CIDP
Record Dates: First submitted 2020-08-21; First posted 2020-08-27 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Chronic Inflammatory Demyelinating Polyradiculoneuropathy
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group with walking disorder (Other): This Group with walking disorder corresponds to patient reporting walking disorders due to his illness.
  Interventions: Other: Group with walking disorder
- Group without walking disorder (Other): This Group without walking disorder corresponds to patients not reporting walking disorders due to his illness.
  Interventions: Other: Group without walking disorder

INTERVENTIONS:
Other: Group with walking disorder — During the patient's hospitalization, two questionnaires will be completed, assessing the handicap of the patient in his daily activities, and the specific incapacity to carry out activities of daily living and social life (10 minutes to complete). The patient will then carry out two 20-meter round-trip walking tests during his first day and his last day of care at the hospital. Additional home visits, corresponding to intervention, performed by a member of the investigative team, will take place once a week (15-20 minutes). The team will collect his feelings about the evolution of symptoms through the two questionnaires, and quantify the evolution of his walking. Walk tests are recorded using small inertial sensors (accelerometers and gyrometers) that will be placed at his feet, belt and forehead. This examination is not painful. All the measurements are carried out in 15 minutes by a member of the team.
  Arms: Group with walking disorder
Other: Group without walking disorder — During the patient's hospitalization, two questionnaires will be completed, assessing the handicap of the patient in his daily activities, and the specific incapacity to carry out activities of daily living and social life (10 minutes to complete). The patient will then carry out two 20-meter round-trip walking tests during his first day and his last day of care at the hospital.
  Additional home visits, corresponding to interventions, performed by a member of the investigative team, will take place once a week (15-20 minutes). The team will collect his feelings about the evolution of symptoms through the two questionnaires, and quantify the evolution of his walking. Walk tests are recorded using small inertial sensors (accelerometers and gyrometers) that will be placed at his feet, belt and forehead. This examination is not painful. All the measurements are carried out in 15 minutes by a member of the team.
  Arms: Group without walking disorder

SUMMARY:
Chronic inflammatory demyelinating polyradiculoneuropathy is a diffuse multifocal autoimmune disorder of the peripheral neuron, affecting 1 to 9 in 100,000 people. Its course is difficult to predict, and may be characterized by continuous progression, multiple relapses, or recovery after a few months. treatment. The predominantly motor form with 4 limbs represents the typical form, but the disease can take on other clinical forms (pure sensory impairment, ataxia, etc.).

In addition to induction therapy, patients most often require long-term maintenance therapy. First-line therapies, with the same efficacy according to a 2013 Cochrane study, are glucocorticoid therapy, plasma exchanges and intravenous immunoglobulin injections. Glucocorticoids have a grade C recommendation level while a grade A has been assigned to intravenous immunoglobulins and plasma exchange. However, the latter have less tolerance and have a rebound effect which limits their long-term interest. Intravenous immunoglobulins are therefore the preferred treatment today. The effect of intravenous immunoglobulins, delivered as a bolus over a few days, lasts two to six weeks, with the number of people being cured of three to improve a person. A more recent study has also shown their advantage in reducing the relapse rate at 6 months.

However, the response to intravenous immunoglobulins fluctuates in different patients and, for any given patient, changes over the course of the disease. The 2010 recommendations therefore recommend an adaptation of the doses and duration of intercourse (0.4 to 1.2 g / kg every 2 to 6 weeks) according to individual monitoring of the response to treatment. In order to embrace the diversity of symptoms of chronic inflammatory demyelinating polyradiculoneuropathy, several scores and scales are usually combined to ensure this follow-up in a cohort. Three clinical data are currently favored: the Inflammatory Rasch-built Overall Disability Scale (I-RODS), the INCAT Overall Neuropathy Limitations Scale (ONLS), the score of the Medical Research Council (MRC). However, none of them assess walking objectively.

However, patients with chronic inflammatory demyelinating polyradiculoneuropathy sometimes report significant walking disturbances, which may result from both sensory disturbances or motor disturbances present in varying degrees depending on the patient. The alterations concerned, according to the studies, the walking speed, the temporal pattern of the step, with an impairment of the durations of the different phases (support and oscillation) or the angle and the angular speed of roll at the level of the trunk. Alterations in speed and phase duration of the step improve during treatment with intravenous immunoglobulin cures, with greater sensitivity compared to the ONLS and MRC scales. The power of the propulsive moment at the ankle during the last moments of the stance phase - the push-off - is another promising gait parameter that has made it possible to distinguish diabetic patients with polyneuropathy from those without diabetes. polyneuropathy and the intensity of the deficit is linked to the severity of the attack. Gait speed, as a reflection of the subject's gait performance, and the quality of gait including the timing of gait, trunk rotation movements and push-off, therefore seem to be potential response markers. for monitoring patients treated with intravenous immunoglobulins.

InertiaLocoGraphy, quantification of gait by inertial measurement sensors, has proven its value in the evaluation of various pathologies in neurological practice, including chronic inflammatory demyelinating polyradiculoneuropathy. It gives access to the walking speed as well as to various walking quality criteria (vigor of the step, rhythmicity, regularity, symmetry, stability, fluidity, synchronization) including the times of the different walking phases and the rotational movements of the trunk, and a push-off substitute.

InertiaLocoGraphie, non-invasive, easy and quick to set up, reflecting the patient's function, therefore potentially provides biomarkers of choice for monitoring the response to intravenous immunoglobulin cures in patients with chronic inflammatory polyradiculoneuropathy demyelinating. Its association with the traditional monitoring tools such as the ONLS score, the I-ROS, and the CRM therefore appears to be of key interest for this monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is ≥ 18 years
* Patient diagnosed with chronic inflammatory demyelinating polyneuropathy (CIDP) in one of the following two cases:

  * Certain IPDC according to ENFS / PNS 2010 criteria
  * Possible or probable CIDP according to ENFS / PNS 2010 criteria with favorable response to immunomodulatory treatment 23
* Patient treated with IVIG
* Mobile patient, able to walk 2 sets of 20 m with a half turn, with a 3 min break between the two exercises.

Patients will be included in one of the following two groups:

* G_CIDP: if the patient reports walking disorders due to his illness
* NG_CIDP: otherwise

  * Patient living in an area accessible by public transport with a journey time of 1 hour (sector ≈ 5 - 6 km)
  * Patient affiliated to a social security scheme
  * Patient who has given oral, free, informed and express consent

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty
* Pregnant woman
* Patient with a pathology other than IPDC that may affect walking (muscular-skeletal pathology, other neurological pathology, etc.) according to the attached clinical questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-16 (Actual); Primary Completion 2022-04-16 (Actual); Study Completion 2022-04-16 (Actual)

PRIMARY OUTCOMES:
Push-off Variation between D1 and D15 | Day 15
  This outcome corresponds to comparison of the absolute variation of Push-off (corresponding to the power of the moment of propulsion at the ankle during the last moments of the support phase) between D0 and D15 in the three subgroups defined by the change in ONLS at D15.

SECONDARY OUTCOMES:
Push-off Variation at Day 4 | Day 4
  This outcome corresponds to comparison of the absolute variation of Push-off (corresponding to the power of the moment of propulsion at the ankle during the last moments of the support phase) between D0 and D4 in the three subgroups defined by the change in ONLS.
Walking speed Variation at Day 4 | Day 4
  This outcome corresponds to comparison of the absolute variation of the walking speed and the quality criteria of walking (vigor of the step, rhythmicity, regularity, symmetry, stability, fluidity, synchronization) between D0 and D4 in the three sub-groups defined by the change in ONLS on D15 (Subgroups: responders if ONLS decrease by more than 1 point, non-responder if ONLS is stable, progressors if ONLS increase by more than 1 point) in groups of patients with and without walking disorders
Walking speed Variation at Day 15 | Day 15
  This outcome corresponds to comparison of the absolute variation of the walking speed and the quality criteria of walking (vigor of the step, rhythmicity, regularity, symmetry, stability, fluidity, synchronization) between D0 and D15 in the three sub-groups defined by the change in ONLS on D15 (Subgroups: responders if ONLS decrease by more than 1 point, non-responder if ONLS is stable, progressors if ONLS increase by more than 1 point) in groups of patients with and without walking disorders

CONTACTS AND LOCATIONS:
Overall Officials: Pauline REACH, MD, Principal Investigator — Fondation Hôpital Saint-Joseph

REFERENCES:
- [Result] Laughlin RS, Dyck PJ, Melton LJ 3rd, Leibson C, Ransom J, Dyck PJ. Incidence and prevalence of CIDP and the association of diabetes mellitus. Neurology. 2009 Jul 7;73(1):39-45. doi: 10.1212/WNL.0b013e3181aaea47. PMID 19564582
- [Result] Dyck PJ, O'Brien PC, Oviatt KF, Dinapoli RP, Daube JR, Bartleson JD, Mokri B, Swift T, Low PA, Windebank AJ. Prednisone improves chronic inflammatory demyelinating polyradiculoneuropathy more than no treatment. Ann Neurol. 1982 Feb;11(2):136-41. doi: 10.1002/ana.410110205. PMID 7041788
- [Result] Eftimov F, Winer JB, Vermeulen M, de Haan R, van Schaik IN. Intravenous immunoglobulin for chronic inflammatory demyelinating polyradiculoneuropathy. Cochrane Database Syst Rev. 2013 Dec 30;(12):CD001797. doi: 10.1002/14651858.CD001797.pub3. PMID 24379104
- [Result] Van den Bergh PY, Hadden RD, Bouche P, Cornblath DR, Hahn A, Illa I, Koski CL, Leger JM, Nobile-Orazio E, Pollard J, Sommer C, van Doorn PA, van Schaik IN; European Federation of Neurological Societies; Peripheral Nerve Society. European Federation of Neurological Societies/Peripheral Nerve Society guideline on management of chronic inflammatory demyelinating polyradiculoneuropathy: report of a joint task force of the European Federation of Neurological Societies and the Peripheral Nerve Society - first revision. Eur J Neurol. 2010 Mar;17(3):356-63. doi: 10.1111/j.1468-1331.2009.02930.x. PMID 20456730
- [Result] Adrichem ME, Eftimov F, van Schaik IN. Intravenous immunoglobulin treatment in chronic inflammatory demyelinating polyradiculoneuropathy, a time to start and a time to stop. J Peripher Nerv Syst. 2016 Sep;21(3):121-7. doi: 10.1111/jns.12176. PMID 27241239
- [Result] Hughes RA, Donofrio P, Bril V, Dalakas MC, Deng C, Hanna K, Hartung HP, Latov N, Merkies IS, van Doorn PA; ICE Study Group. Intravenous immune globulin (10% caprylate-chromatography purified) for the treatment of chronic inflammatory demyelinating polyradiculoneuropathy (ICE study): a randomised placebo-controlled trial. Lancet Neurol. 2008 Feb;7(2):136-44. doi: 10.1016/S1474-4422(07)70329-0. PMID 18178525
- [Result] Kuitwaard K, van Doorn PA. Newer therapeutic options for chronic inflammatory demyelinating polyradiculoneuropathy. Drugs. 2009 May 29;69(8):987-1001. doi: 10.2165/00003495-200969080-00004. PMID 19496628
- [Result] Debs R, Reach P, Cret C, Demeret S, Saheb S, Maisonobe T, Viala K. A new treatment regimen with high-dose and fractioned immunoglobulin in a special subgroup of severe and dependent CIDP patients. Int J Neurosci. 2017 Oct;127(10):864-872. doi: 10.1080/00207454.2016.1269328. Epub 2016 Dec 20. PMID 27918219
- [Result] Oudre L, Barrois-Muller R, Moreau T, Truong C, Vienne-Jumeau A, Ricard D, Vayatis N, Vidal PP. Template-Based Step Detection with Inertial Measurement Units. Sensors (Basel). 2018 Nov 19;18(11):4033. doi: 10.3390/s18114033. PMID 30463240
- [Result] Antoine JC, Azulay JP, Bouche P, Creange A, Fournier E, Gallouedec G, Lagueny A, Lefaucheur JP, Leger JM, Magy L, Maisonobe T, Nicolas G, Pouget J, Soichot P, Stojkovic T, Vallat JM, Verschueren A, Vial C, Viala K; Groupe d'Etude francais des PIDC. [Chronic inflammatory demyelinating polyradiculoneuropathy: diagnostic strategy. Guidelines of the French CIDP study group]. Rev Neurol (Paris). 2005 Oct;161(10):988-96. doi: 10.1016/s0035-3787(05)85166-5. French. PMID 16365632
- [Result] Vienne A, Barrois RP, Buffat S, Ricard D, Vidal PP. Inertial Sensors to Assess Gait Quality in Patients with Neurological Disorders: A Systematic Review of Technical and Analytical Challenges. Front Psychol. 2017 May 18;8:817. doi: 10.3389/fpsyg.2017.00817. eCollection 2017. PMID 28572784
- [Result] Vienne-Jumeau A, Oudre L, Moreau A, Quijoux F, Edmond S, Dandrieux M, Legendre E, Vidal PP, Ricard D. Personalized Template-Based Step Detection From Inertial Measurement Units Signals in Multiple Sclerosis. Front Neurol. 2020 Apr 21;11:261. doi: 10.3389/fneur.2020.00261. eCollection 2020. PMID 32373047
- [Result] Andersen H, Jakobsen J. A comparative study of isokinetic dynamometry and manual muscle testing of ankle dorsal and plantar flexors and knee extensors and flexors. Eur Neurol. 1997;37(4):239-42. doi: 10.1159/000117450. PMID 9208265
- [Result] Rao S, Saltzman C, Yack HJ. Ankle ROM and stiffness measured at rest and during gait in individuals with and without diabetic sensory neuropathy. Gait Posture. 2006 Nov;24(3):295-301. doi: 10.1016/j.gaitpost.2005.10.004. Epub 2005 Nov 15. PMID 16293415